CLINICAL TRIAL: NCT03055884
Title: Investigating Accelerated Learning in Healthy Subjects
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: low numbers of participants
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Sven Vanneste, Associate professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-34
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-04

CONDITIONS: Healthy Adults
Keywords: transcranial Direct Current Stimulation (tDCS); accelerated learning; memory
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- active tDCS with repeated retrieval practice (Experimental): active tDCS with verbal paired-associate learning task with repeated retrieval practice
  Interventions: Device: tDCS; Behavioral: Verbal paired-associate learning task
- active tDCS without repeated retrieval practice (Experimental): active tDCS with verbal paired-associate learning task without repeated retrieval practice
  Interventions: Device: tDCS; Behavioral: Verbal paired-associate learning task
- Sham tDCS with repeated retrieval practice (Sham Comparator): sham tDCS with verbal paired-associate learning task with repeated retrieval practice
  Interventions: Behavioral: Verbal paired-associate learning task
- Sham tDCS without repeated retrieval practice (Sham Comparator): shamtDCS with verbal paired-associate learning task without repeated retrieval practice
  Interventions: Behavioral: Verbal paired-associate learning task

INTERVENTIONS:
Device: tDCS — active tDCS versus sham tDCS
  Arms: active tDCS with repeated retrieval practice; active tDCS without repeated retrieval practice
Behavioral: Verbal paired-associate learning task — with or without repeated retrieval practice

SUMMARY:
The purpose of this study is to investigate whether it is possible to accelerate learning and improve associative memory performance in healthy subjects, by (1) applying transcranial Direct Current Stimulation (tDCS) during a verbal paired-associate learning task and by (2) optimizing the learning method with repeated retrieval practice.

DETAILED DESCRIPTION:
Associative memory refers to remembering the association between two items, such as a face and a name or a word in English and the same word in another language. It is not only important for learning, but it is also one of the first aspects of memory performance that is impacted by aging and by Alzheimer׳s disease. For decades, neuroscientists have investigated associative learning and memory and ways to accelerate and enhance associative learning and memory.

Transcranial Direct Current stimulation (tDCS) is a non-invasive and painless electrical stimulation technique that has demonstrated to accelerate learning and improve memory in some studies. Previous research has also emphasized the importance of repeated retrieval practice as a way to accelerate learning and enhance associative memory performance. Therefore, this study will examine the effect of repeated retrieval practice on associative memory performance by using two versions of an associative memory task.

To investigate whether it is possible to accelerate learning and improve associative memory using tDCS and repeated retrieval practice, the performance in a Verbal Paired-Associate memory task during the first visit and 1 week after will be compared for four study groups. The first group will get active tDCS during a version of the verbal paired-associate learning task with repeated retrieval practice. The second group will get active tDCS during a version of the verbal paired-associate learning task without repeated retrieval practice. The third group will get sham tDCS during a version of the verbal paired-associate learning task with repeated retrieval practice and the fourth group will get Sham tDCS during a version of the verbal paired-associate learning task without repeated retrieval practice.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 years
* Native English Speaker

Exclusion Criteria:

* History of severe head injuries,epileptic insults, or heart disease
* Severe psychiatric disorders and severe untreated medical problems.
* Acquainted with the foreign language used in the learning task
* Contraindications for tDCS (pregnant women, implanted devices)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2021-12-22 (Estimated)

PRIMARY OUTCOMES:
Associative Memory assessed by a Verbal Paired-Associate memory test | baseline and 1 week after the tDCS
  Changes in performance in the Verbal Paired-Associate memory task is compared between the 4 groups (1. tDCS+verbal paired-associate learning task with repeated retrieval practice, 2. tDCS + verbal paired-associate learning task without repeated retrieval practice, 3. Sham tDCS+verbal paired-associate learning task with repeated retrieval practice, 4. Sham tDCS + verbal paired-associate learning task without repeated retrieval practice) to investigate the influence of tDCS and learning method on Associative Memory

CONTACTS AND LOCATIONS:
Overall Officials: Sven Vanneste, Principal Investigator — The University of Texas at Dallas
Locations (1):
- The University of Texas of Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided